CLINICAL TRIAL: NCT03443635
Title: Cooking for Health Optimization With Patients
Acronym: CHOP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHOP
Record Dates: First submitted 2018-02-10; First posted 2018-02-23 (Actual); Results first posted 2022-02-25 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; Nutrition Disorders; Diabetes; Hypertension; Cancer; Depression; Obesity; Physical Activity
MeSH Terms: conditions — Cardiovascular Diseases; Nutrition Disorders; Diabetes Mellitus; Hypertension; Neoplasms; Depression; Obesity; Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Subjects receiving hands-on cooking and nutrition education classes
  Interventions: Behavioral: Treatment
- Control (No Intervention): Subjects not receiving any additional nutrition education aside from that contained in their curricula (for trainees) or medical care (for patients)

INTERVENTIONS:
Behavioral: Treatment — The intervention educates subjects through the hands-on cooking and nutrition education classes how to buy, cook, store, and consume healthy foods as an adjunct to healthy activity levels and avoidance of such health risks factors as smoking, excessive alcohol intake, and drug use.
  Arms: Treatment

SUMMARY:
Cooking for Health Optimization with Patients (CHOP) is the first known multi-site prospective cohort study with a nested Bayesian adaptive randomized trial in the preventive cardiology field of culinary medicine. It is also the first known longitudinal study to assess the impact of hands-on cooking and nutrition education on patient outcomes, with those classes taught by medical students and other future and current medical professionals who have first been trained in those classes on how to integrate diet and lifestyle counseling of patients with their respective scopes of clinical practice. CHOP is the primary research study of the world's first known medical school based teaching kitchen, The Goldring Center for Culinary Medicine at Tulane University School of Medicine. Medical trainees and professionals are followed in this study long-term to understand how the classes impact their competencies in patient counseling, attitudes about the counseling, and their own diets. Patients who consent to being randomized to these classes compared to standard of care are studied within the nested Bayesian adaptive randomized trial to understand how the classes impact their health outcomes, clinical and food costs, and the costs of health systems caring for these patient populations. CHOP is designed as a pragmatic population health trial to hopefully improve healthcare effectiveness, equity, and cost by establishing an evidence-based, scalable, sustainable model of healthcare intervention targeting the social determinants of health, while complementing the pharmacological and/or surgical management of patients.

ELIGIBILITY:
Inclusion Criteria:

* 7 to 115 years of age (patients), and currently a medical trainee or professional (including for physicians, nurses, physician assistants, and dieticians)

Exclusion Criteria:

* Inability to complete at least 2 intervention classes

Ages: 7 Years to 115 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7192 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Monlezun, MD, PhD, MPH, Principal Investigator — The Goldring Center for Culinary Medicine at Tulane University School of Medicine
Locations (1):
- The Goldring Center for Culinary Medicine at Tulane University School of Medicine, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monlezun DJ, Kasprowicz E, Tosh KW, Nix J, Urday P, Tice D, Sarris L, Harlan TS. Medical school-based teaching kitchen improves HbA1c, blood pressure, and cholesterol for patients with type 2 diabetes: Results from a novel randomized controlled trial. Diabetes Res Clin Pract. 2015 Aug;109(2):420-6. doi: 10.1016/j.diabres.2015.05.007. Epub 2015 May 12. PMID 26002686
- [Background] Monlezun DJ, Leong B, Joo E, Birkhead AG, Sarris L, Harlan TS. Novel Longitudinal and Propensity Score Matched Analysis of Hands-On Cooking and Nutrition Education versus Traditional Clinical Education among 627 Medical Students. Adv Prev Med. 2015;2015:656780. doi: 10.1155/2015/656780. Epub 2015 Sep 8. PMID 26435851
- [Background] Monlezun DJ, Carr C, Niu T, Nordio F, DeValle N, Sarris L, Harlan T. Meta-analysis and machine learning-augmented mixed effects cohort analysis of improved diets among 5847 medical trainees, providers and patients. Public Health Nutr. 2022 Feb;25(2):281-289. doi: 10.1017/S1368980021002809. Epub 2021 Jun 28. PMID 34176552
- [Background] Razavi AC, Sapin A, Monlezun DJ, McCormack IG, Latoff A, Pedroza K, McCullough C, Sarris L, Schlag E, Dyer A, Harlan TS. Effect of culinary education curriculum on Mediterranean diet adherence and food cost savings in families: a randomised controlled trial. Public Health Nutr. 2021 Jun;24(8):2297-2303. doi: 10.1017/S1368980020002256. Epub 2020 Aug 3. PMID 32744215
- [Background] Patnaik A, Tran J, McWhorter JW, Burks H, Ngo A, Nguyen TD, Mody A, Moore L, Hoelscher DM, Dyer A, Sarris L, Harlan T, Chassay CM, Monlezun D. Regional variations in medical trainee diet and nutrition counseling competencies: Machine learning-augmented propensity score analysis of a prospective multi-site cohort study. Med Sci Educ. 2020 May 20;30(2):911-915. doi: 10.1007/s40670-020-00973-6. eCollection 2020 Jun. PMID 34457749
- [Background] Razavi AC, Monlezun DJ, Sapin A, Stauber Z, Schradle K, Schlag E, Dyer A, Gagen B, McCormack IG, Akhiwu O, Sarris L, Dotson K, Harlan TS. Multisite Culinary Medicine Curriculum Is Associated With Cardioprotective Dietary Patterns and Lifestyle Medicine Competencies Among Medical Trainees. Am J Lifestyle Med. 2020 Jan 24;14(2):225-233. doi: 10.1177/1559827619901104. eCollection 2020 Mar-Apr. PMID 32231488
- [Background] Razavi AC, Monlezun DJ, Sapin A, Sarris L, Schlag E, Dyer A, Harlan T. Etiological Role of Diet in 30-Day Readmissions for Heart Failure: Implications for Reducing Heart Failure-Associated Costs via Culinary Medicine. Am J Lifestyle Med. 2019 Jul 14;14(4):351-360. doi: 10.1177/1559827619861933. eCollection 2020 Jul-Aug. PMID 33281513
- [Background] Wetherill MS, Davis GC, Kezbers K, Carter V, Wells E, Williams MB, Ijams SD, Monlezun D, Harlan T, Whelan LJ. Development and Evaluation of a Nutrition-Centered Lifestyle Medicine Curriculum for Physician Assistant Students. Med Sci Educ. 2018 Dec 6;29(1):163-172. doi: 10.1007/s40670-018-00655-4. eCollection 2019 Mar. PMID 34457464
- [Background] Monlezun DJ, Dart L, Vanbeber A, Smith-Barbaro P, Costilla V, Samuel C, Terregino CA, Abali EE, Dollinger B, Baumgartner N, Kramer N, Seelochan A, Taher S, Deutchman M, Evans M, Ellis RB, Oyola S, Maker-Clark G, Dreibelbis T, Budnick I, Tran D, DeValle N, Shepard R, Chow E, Petrin C, Razavi A, McGowan C, Grant A, Bird M, Carry C, McGowan G, McCullough C, Berman CM, Dotson K, Niu T, Sarris L, Harlan TS, Co-Investigators OBOTC. Machine Learning-Augmented Propensity Score-Adjusted Multilevel Mixed Effects Panel Analysis of Hands-On Cooking and Nutrition Education versus Traditional Curriculum for Medical Students as Preventive Cardiology: Multisite Cohort Study of 3,248 Trainees over 5 Years. Biomed Res Int. 2018 Apr 15;2018:5051289. doi: 10.1155/2018/5051289. eCollection 2018. PMID 29850526
- [Background] Kasprowicz E, Monlezun DJ, Harlan TS. Letter by Kasprowicz et al regarding article, "reducing sodium intake to prevent stroke: time for action, not hesitation". Stroke. 2014 Jun;45(6):e108. doi: 10.1161/STROKEAHA.114.005157. Epub 2014 May 6. No abstract available. PMID 24803593
- [Background] Birkhead AG, Foote S, Monlezun DJ, Loyd J, Joo E, Leong B, Sarris L, Harlan TS. Medical student-led community cooking classes: a novel preventive medicine model that's easy to swallow. Am J Prev Med. 2014 Mar;46(3):e41-2. doi: 10.1016/j.amepre.2013.11.006. No abstract available. PMID 24512876
- See also: Related Info — http://culinarymedicine.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 2616 | 4576
Completed | 2127 | 3720
Not Completed | 489 | 856

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 2616 | 4576 | 7192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1870 | 3571 | 5441
  >=65 years | 746 | 1005 | 1751
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.02 (12.69) | 28.16 (8.48) | 29.49 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1700 | 2725 | 4425
  Male | 916 | 1851 | 2767
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 39 | 14 | 53
  Asian | 376 | 709 | 1085
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 556 | 507 | 1063
  White | 1262 | 2601 | 3863
  More than one race | 383 | 745 | 1128
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2616 | 4576 | 7192

OUTCOME MEASURES:

1. Primary Outcome: High or Medium (Versus Low) Mediterranean Diet Adherence
Description: Based on 9-point Trichopoulou et al. 2003 NEJM scale (for patients, medical trainees, and providers)
Time Frame: 6 months
Measure: Number; unit: percentage of arm
Groups:
- Control: Subjects not receiving any additional nutrition education aside from that contained in their curricula (for trainees/providers) or medical care (for patients)
Arm/Group | Treatment | Control
Number analyzed (Participants) | 2616 | 4576
percentage of arm | 55.99 | 50.53

2. Secondary Outcome: Hospital Readmissions
Description: Re-presenting to the hospital for similar presenting diagnosis (for patients)
Time Frame: 30 days
Reporting Status: Not Posted

3. Secondary Outcome: Composite Rate of All Cause-mortality, Myocardial Infarction, and Cerebrovascular Event
Description: (For patients)
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Competencies
Description: Educating patients on healthy diet and lifestyles according to 25 competency topics (for medical trainees)
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Healthcare Costs
Description: Direct and indirect (for patients)
Time Frame: 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Healthcare Costs
Description: Direct and indirect (for health systems caring for the patients in the trial)
Time Frame: 6 months
Reporting Status: Not Posted

7. Secondary Outcome: Food Costs
Description: Grocery and restaurant costs (for patients)
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/2616 | 0/4576
Serious Adverse Events (participants affected / at risk) | 0/2616 | 0/4576
Other Adverse Events (participants affected / at risk) | 0/2616 | 0/4576

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT03443635/Prot_SAP_000.pdf